CLINICAL TRIAL: NCT03884010
Title: Accuracy of Anthropometric Equations to Estimate DXA-Derived Skeletal Muscle Mass in Professional Male Soccer Players
Status: Completed | Type: Observational
Sponsor: Centro Universitario de Ciencias de la Salud, Mexico (Other)
Responsible Party: Principal Investigator, Juan Ricardo Lopez y Taylor, Director of the Institute of Applied Sciences for Physical Activity and Sport, Centro Universitario de Ciencias de la Salud, Mexico
Other Study IDs: LNFUT-2
Record Dates: First submitted 2019-03-19; First posted 2019-03-21 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Body Composition
Keywords: DXA; Soccer players; Skeletal muscle mass

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Professional male soccer players from the second professional Mexican division
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Cross-sectional

SUMMARY:
This study aimed to analyze the accuracy of different anthropometric equations to estimate skeletal muscle mass in professional male soccer players, setting dual-energy x-ray absorptiometry (DXA) skeletal muscle mass as the reference.

DETAILED DESCRIPTION:
The study consisted of evaluating anthropometric measurements and body composition with DXA in professional male soccer player aged 18 years and older. Standardized and certified personnel carried out anthropometric measurements and DXA whole body scan the same day.

Skeletal muscle mass was estimated with several anthropometric equations. The reference skeletal muscle mass was obtained assessing appendicular lean soft tissue from a whole-body DXA scan and then transformed into skeletal muscle mass with Kim equation (2002).

The estimated skeletal muscle mass from anthropometric equations was compared with DXA, and those with non-significant differences were further analyzed for calculating mean differences and 95% limits of agreement with DXA. This analysis was carried out for all equations.

ELIGIBILITY:
Inclusion Criteria:

* Signed contract with the team

Exclusion Criteria:

* Injured

Ages: 18 Years to 37 Years | Sex: Male
Age Groups: Adult
Study Population: Professional male soccer players hired into a second professional Mexican division team.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle mass | One day
  Skeletal muscle mass was obtained from assessing appendicular lean soft tissue from a DXA whole body scan, and then transformed into skeletal muscle mass with Kim equation (2002).

CONTACTS AND LOCATIONS:
Overall Officials: Juan R López-Taylor, Study Director — University of Guadalajara
Locations (1):
- Instituto de Ciencias Aplicadas a la Actividad Física y al Deporte, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Undecided